CLINICAL TRIAL: NCT06241547
Title: Perioperative Percutaneous Electrical Nerve Stimulation Via a Wearable Equipment on Postoperative Nausea and Vomiting（PONV） in Patients Undergoing Laparoscopy Abdominal Surgery: a Prospective Randomized Controlled Trial
Brief Title: PONV Prevention Via Percutaneous Nerve Electrical Stimulation on PC6
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: I-23PJ1712
Record Dates: First submitted 2023-10-31; First posted 2024-02-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimulation group (Experimental): accept general drug prevention, wear the equipment, and receive electrical stimulation.
  Interventions: Device: electrical stimualtion via EmeTerm bracelet; Drug: antimetic drugs（ dexamethasone，ondansetron）
- control group (Placebo Comparator): accept general drug prevention and wear the equipment but receive no electrical stimulation
  Interventions: Drug: antimetic drugs（ dexamethasone，ondansetron）

INTERVENTIONS:
Device: electrical stimualtion via EmeTerm bracelet — We planned to exert electrical stimulation via the bracelet.
  Arms: stimulation group
Drug: antimetic drugs（ dexamethasone，ondansetron） — Antimetic drugs (dexamethasone ondansetron) are used to prevent postoperative nausea and vomiting.

SUMMARY:
This study aims to certify the effectiveness of percutaneous electrical nerve stimulation at Pericardium 6 (PC6) via a wearable equipment during perioperative period on preventing postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Introduction: This study aims to certify the effectiveness of percutaneous electrical nerve stimulation at Pericardium 6 (PC6) via a wearable equipment during perioperative period on preventing postoperative nausea and vomiting.

Method and analysis: A total of approximately 302 patients undergoing elective laparoscopic surgery will be enrolled. Participants will be randomly assigned to either a electrical stimulation group or a placebo group, with computer-generated randomization and concealed allocation using sealed envelopes. The electrical stimulation group will receive PC point electrical stimulation 30 minutes before surgery until 24 hours postoperatively, while the placebo group will wear a wristband without stimulation. The primary outcome will be the incidence of postoperative nausea and vomiting, with secondary outcomes including the incidence of nausea and vomiting within 24 hours after surgery, gastrointestinal and hemodynamic indices, postoperative recovery, hospital stay and cost, and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years;
2. Patients undergoing elective laparoscopic surgery;
3. American Society of Anaesthesiologists(ASA) Grade 1 to 3;
4. Anesthesia: General Anesthesia, Tracheal Intubation;
5. BMI: ≥18, <28;
6. Gender: female
7. Patients or their family members are able to comprehend the study protocol and are willing to participate in this research by providing written informed consent.

Exclusion Criteria:

1. There are incisions or scars in the wearing position of the device;
2. There is a local infection in the wearing position of the device;
3. upper extremity nerve injury;
4. history of spinal cord surgery;
5. Participated in other clinical trials within 4 weeks;
6. suffering from severe central nervous system disease or mental disorder;
7. Patients need to return to the ICU after surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting(PONV) | 24 hours after surgery
  Ask patients if they experienced nausea or vomiting 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Response:
  Thank you for your comment. We plan to share Individual Participant Data (IPD) upon request. Researchers interested in accessing the data can contact the corresponding author via email. The data will be shared following a review of the request to ensure that it complies with ethical guidelines and protects participant privacy.
Supporting Information: Study Protocol, CSR
Time Frame: 5 years after study completion
Access Criteria: e-mail to tracymaobao@126.com

REFERENCES:
- [Derived] Chen J, Che L, Cui Q, Lang J, Zhang Y, Zhu B, Huang Y. Acustimulation combined with pharmacological prophylaxis versus pharmacological prophylaxis alone in postoperative nausea and vomiting (PONV) prophylaxis among patients undergoing laparoscopy abdominal surgery: a research protocol for a randomised controlled trial. BMJ Open. 2024 Sep 23;14(9):e088633. doi: 10.1136/bmjopen-2024-088633. PMID 39313286